CLINICAL TRIAL: NCT02806648
Title: A Phase II Trial to Assess the Activity and Safety of Palbociclib in Patients With Well and Moderately Differentiated Metastatic Pancreatic Neuroendocrine Tumors (pNET)
Brief Title: A Trial to Assess the Activity and Safety of Palbociclib in Patients With Well and Moderately Differentiated Metastatic Pancreatic Neuroendocrine Tumors (pNET)
Acronym: PALBONET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Espanol de Tumores Neuroendocrinos (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GETNE-1407
Record Dates: First submitted 2015-07-08; First posted 2016-06-20 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2016-06

CONDITIONS: Pancreatic Neuroendocrine Cancer
MeSH Terms: conditions — Somatostatinoma | interventions — palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Palbociclib (Experimental): Palbociclib
  Interventions: Drug: Palbociclib

INTERVENTIONS:
Drug: Palbociclib — Palbociclib
  Other Names: palbociclib (PD0332991)

SUMMARY:
A phase II trial to assess the activity and safety of PD0332991 in patients with well- and moderately-differentiated metastatic pancreatic neuroendocrine tumors (pNET) with overexpression of cell cycle markers (Cdk4 and/or phospho-Rb1 and/or cyclin D1)

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the activity and safety of PD0332991 in patients with well- and moderately-differentiated metastatic pancreatic neuroendocrine tumors (pNET) with overexpression of cell cycle markers (Cdk4 and/or phospho-Rb1 and/or cyclin D1)

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically proven diagnosis of pancreatic neuroendocrine tumors (pNET) with Ki67 assessment of < or = 20% (well and moderately differentiated) with evidence of unresectable disease or metastatic disease. Locally advanced disease must not be amendable to resection or radiation therapy with curative intent.
2. Overexpression of Cdk4 and/or phospho-Rb1 and/or cyclin D1 in tumor tissue sample from tumor biopsy or prior primary tumor resection (Molecular study will be conducted at CNIO and logistic is described later). Therefore availability of paraffin-embedding tumor tissue sample is needed.
3. Documented progression of the disease by CT scan, MRI, or Octreoscan within 12 months prior to baseline.
4. Previous treatments with chemotherapy, antiangiogenics, or interferon are permitted providing that toxicity has resolved to < grade 1 at study entry and that last treatment was at least 4 weeks prior to baseline assessment. Patients may be treated with somatostatin analogues during the trial. Concomitant interferon treatment is not permitted.
5. Measurable disease as per RECIST. Measurable lesions that have been previously radiated will not be considered target lesions unless increase in size has been observed following completion of radiation therapy.
6. Able to swallow oral compound
7. Male or female, 18 years of age or older.
8. ECOG performance status less than 2.
9. Life expectancy greater than 12 weeks.
10. The definitions of minimum adequacy for organ function required prior to study entry are as follows. In addition, safety precautions provided in the product labeling for the anticipated control arm chemotherapy must be observed.

    * Serum aspartate transaminase (AST) and serum alanine transaminase (ALT) 2.5 x upper limit of normal (ULN), or AST and ALT 5 x ULN if liver function abnormalities are due to underlying malignancy
    * Total serum bilirubin 1.5 x ULN
    * Serum albumin 3.0 g/dL
    * Absolute neutrophil count (ANC) 1500/L
    * Platelets 100,000/L
    * Hemoglobin 9.0 g/dL
    * Creatinin clearance < 40 mL/min
11. Signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all the pertinent aspects of the trial prior to enrollment.
12. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Prior chemotherapy regimen or biological treatment for locally advanced or metastatic transitional cell carcinoma of the urinary tract.
2. Prior treatment on Cdk4 inhibitor under clinical trial.
3. Creatinine clearance < 40 ml/min using Cockroft and Gault formula.
4. Major surgery, radiation therapy, or systemic therapy within 3 weeks of study randomization except palliative radiotherapy to non-target metastatic lesions.
5. Prior high-dose chemotherapy requiring hematopoietic stem cell rescue.
6. Immunosuppressive drugs such as cyclosporine, tacrolimus, azathioprine, or long-term oral glucocorticoids taken concurrently or within last 3 months prior to randomization
7. Prior radiation therapy to >25% of the bone marrow.
8. Current treatment on another clinical trial.
9. Uncontrolled brain metastases, spinal cord compression, carcinomatous meningitis, or leptomeningeal disease. Patients should have completed surgery or radiation therapy for existing brain metastases, should not have documented increase in size over the previous 3 months prior to first dose of treatment on study and should be asymptomatic.
10. Diagnosis of any second malignancy within the last 3 years, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the cervix.
11. Any of the following within the 12 months prior to starting study treatment: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, congestive heart failure, cerebrovascular accident including transient ischemic attack, or pulmonary embolus.
12. Ongoing cardiac dysrhythmias of NCI CTCAE grade 2, atrial XML File Identifier: 3xAP+CVEwV9UnEoC7xvloFQA/XQ=Page 20/34 fibrillation of any grade, or QTc interval >450 msec for males or >470msec for females.
13. Hypertension that cannot be controlled by medications (>150/100mmHg despite optimal medical therapy)
14. Current treatment with therapeutic doses of Coumadin (low dose Coumadin up to 2 mg PO daily for deep vein thrombosis prophylaxis is allowed).
15. Known human immunodeficiency virus infection.
16. Pregnancy or breastfeeding. All female patients with reproductive potential must have a negative pregnancy test (serum or urine) prior to randomization.
17. Other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that would impart, in the judgment of the investigator, excess risk associated with study participation or study drug administration, or which, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-05; Primary Completion 2017-07 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Activity of palbociclib (PD0332991) considering objective response rate | 20 months

SECONDARY OUTCOMES:
Progression Free Survival | Patients will be followed until disease progression, estimating around 12months
Time to Tumor Progression | Patients will be followed until disease progression, estimating around 12 months
Duration of response | Patients will be followed until disease progression, estimating around 12 months
Overall Survival | Patients will be followed until death, estimating around 33 months
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 (Safety) | Patients will be followed until disease progression estimating around 12 months
  Safety would be measured as Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
Positive expression of tumor biomarkers (Cdk4, Cdk6, fosfo-Rb1, D1 cyclin, p53, Ki67) | Positive expression of tumor biomarkers at baseline
  Percentage of neoplasique cells with positive expression of the following tumor biomarkers Cdk4, Cdk6, fosfo-Rb1, D1 cyclin, p53, Ki67 would be measured at baseline by immunohistochemistry

CONTACTS AND LOCATIONS:
Locations (9):
- Spain (9):
  - ICO, L'Hospitalet de Llobregat, Barcelona
  - C. H. de Navarra, Pamplona, Navarre
  - H.U.C de Asturias, Oviedo, Principality of Asturias
  - H. Vall d´Hebron, Barcelona
  - H. Castellon, Castelló
  - H U Ramón y Cajal, Madrid
  - H. 12 Octubre, Madrid
  - H.U.La Paz, Madrid
  - H.U.Virgen del Rocio, Seville